CLINICAL TRIAL: NCT04014764
Title: An Observational Study to Collect and Assess Tissue Samples From Subjects With One of Three Neoplastic Conditions (ANSWer)
Brief Title: Collect and Assess Tissue Samples From Subjects With Hematologic Malignancy
Acronym: (ANSWer)
Status: Completed | Type: Observational
Sponsor: Notable Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: N-01
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Acute Myelogenous Leukemia; Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The study will require tissue samples taken from consented subjects to be assayed using Notable's ex vivo, high-throughput flow cytometry based platform. The result of this assay will be compared to the subject's documented diagnosis as well as clinical outcome, where applicable. Additional biomarker testing, such as sequencing to determine somatic mutations using targeted panels, may also be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Documented hematologic malignancy in need of starting an active anti-cancer therapy.
  This is a non-interventional study.
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — N/A. This is a non-interventional study. Following consent, the subject will have biospecimen samples taken during routine standard of care procedures, and provided to Sponsor for analysis. Optional research blood draws may occur at treating physician's discretion to obtain additional tissue samples.

SUMMARY:
This is a prospective, multicenter observational study to collect clinically annotated biospecimens in order to assess the correlation between ex vivo data generated by the Notable assay platform and clinical outcome.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational study with collection of de-identified biospecimens with matched clinical data from up to 1000 participants from clinical networks in the United States and Canada. Clinical information, demographics, and medical data relevant to cancer status are collected from all participants and their medical record at baseline (at study entry and time of baseline biospecimen collection), and subsequent visits per patient consent, for up to 1 year.

The primary assessment is the establishment of a tumor registry with annotated clinical outcomes. Exploratory assessments include correlation of ex vivo functional testing results with clinical outcomes, as well as identification of potential biomarkers that correlate responses with genotype and/or phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Age ≥ 18 years, male or female, of any race;
* Documented hematologic malignancy (any of the below) in need of starting an active anti-cancer therapy:
* Acute myelogenous leukemia (AML)
* Multiple myeloma (MM)
* Myelodysplastic syndrome (MDS)
* Lymphoma
* Acute lymphocytic leukemia (ALL)
* Chronic lymphocytic leukemia (CLL)
* Chronic myelogenous leukemia (CML)
* Neoplasm (MPN)
* Other (upon review and approval by medical monitor)

Note: *Supportive care agents including erythropoiesis-stimulating agents (ESAs) such as EPO, Procrit, Aranesp, etc; granulocyte colony stimulating factor (G-CSF); hydroxyurea (Hydrea); and luspatercept (Reblozyl) are not considered anti-cancer therapy for this study

* Intent to start anti-cancer therapy within 21 days of biospecimen collection

  •≥7 days from last anti-cancer therapy;
* Any number of prior therapies
* Subject cohort is currently open

Exclusion Criteria:

* Unwilling or unable to give consent
* Subject's disease is in remission
* Subject cohort is not open at time of consent
* Subject is restarting an ongoing treatment regimen after a dose interruption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1000 Subjects with diagnosed with a hematological malignancy will be enrolled to provide at least 1000 biospecimen samples.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical response to treatment | 3 years
  Collect clinical responses to treatment and outcomes in patients who have provided samples to the biobank

SECONDARY OUTCOMES:
Type of clinical treatment responses | 3 years
  Correlate ex vivo drug sensitivity data on patient samples with clinical treatment responses.
Types of somatic tumor mutations | 3 years
  Determine genotype and/or phenotype relationships between ex vivo and clinical responses with somatic tumor mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroomi Tada, MD, Ph.D., Principal Investigator — Notable Labs
Locations (20):
- United States (11):
  - CBCC Global Research, Bakersfield, California
  - Pacific Central Coast Health Centers -- SLO Oncology and Hematology Health Center, San Luis Obispo, California
  - Colorado West Healthcare System, dba Grand Valley Oncology, Grand Junction, Colorado
  - Ocala Oncology Center, Ocala, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Touro Infirmary, New Orleans, Louisiana
  - Northern Light Cancer Care Center, Brewer, Maine
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - East Carolina University, Greenville, North Carolina
  - The Lindner Center for Research and Education at The Christ Hospital -- The Cancer Center, Cincinnati, Ohio
  - Utah Cancer Specialists, Salt Lake City, Utah
- Greece (6):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - National Kapodistrian University of Athens, Athens
  - Attikon University Hospital, Athens
  - National Kapodistrian Hospital/Laikon General Hospital, Athens
  - University Hospital of Ioánnina, Ioannina
  - University Hospital Patras, Pátrai
- Spain (3):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital San Pedro de Alcántare, Cáceres
  - Hospital Universitari I Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No